CLINICAL TRIAL: NCT00139295
Title: Comparison of the Efficacy and Safety of Hylastan to Methylprednisolone Acetate in Patients With Symptomatic Osteoarthritis of the Knee
Brief Title: Comparison of Hylastan to Methylprednisolone Acetate in Patients With Symptomatic Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVS00103
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Osteoarthritis, Knee
Keywords: musculoskeletal; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee

INTERVENTIONS:
Device: Hylastan

SUMMARY:
This is a clinical study to investigate the safety and efficacy of hylastan in treating patients with symptomatic osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OA of the knee
* Have tried but not been sufficiently helped by conservative treatment, such as weight reduction and pain medications

Exclusion Criteria:

* Prior or concomitant treatments that would impede measurement of safety and efficacy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (24):
- United States (15):
  - Capstone Clinical Trials, Inc, Birmingham, Alabama
  - Hope Research Institute, LLC, Phoenix, Arizona
  - Tucson Orthopedic Institute, PC, Tucson, Arizona
  - Orthopaedic Specialties of Tampa Bay, Clearwater, Florida
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Midwest Orthopedics at Rush University Medical Center, Chicago, Illinois
  - Rockford Health Physicians, Rockford, Illinois
  - Bluegrass Orthopaedics/Bluegrass Musculoskeletal Research, Lexington, Kentucky
  - Orthopedic Specialists of Louisiana, Shreveport, Louisiana
  - Arthritis & Osteoporosis Center of Maryland, Frederick, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Orthopedic Center for Joint Replacement and Sports, Grants Pass, Oregon
  - Coastal Orthopedic Associates, Conway, South Carolina
  - Unlimited Research, San Antonio, Texas
  - Arthritis Northwest, Seattle, Washington
- Sir William Osler Health Institute, Hamilton, Ontario, Canada
- France (3):
  - Clinique du Sport, Mérignac
  - Centre Hospitalier Lyon-Sud, Service de Rhumatologie, Pierre-Bénite
  - CHU Hôpital Trousseau Service de Rhumatologie, Tours
- Germany (2):
  - St-Elisabeth Klinik, Orthopädisch Gemeinschaftspraxis, Heidelberg
  - Orthopaedische Gemeinschaftspraxis, Weyhe-Kirchweyhe
- United Kingdom (3):
  - Southampton General Hospital, MRC Environmental Epidemiology Unit, Southampton, Hampshire
  - Maidstone General Hospital & Tunbridge Wells NHS Trust, Maidstone, Kent
  - Whipps Cross University Hospital NHS Trust, Arthritis Assessment, Physiotherapy Department, Leytonstone, London